CLINICAL TRIAL: NCT03037463
Title: Identification of Tear Biomarkers for Parkinson's Disease Patients
Brief Title: Measuring Parkinson's Disease With Tear Fluid
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sarah Hamm-Alvarez, Professor and Vice Chair, Basic Research; Associate Dean, Basic and Translational Research; Director, Research development, University of Southern California
Other Study IDs: 11594
Record Dates: First submitted 2017-01-12; First posted 2017-01-31 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Parkinson's Disease
- Control

SUMMARY:
The purpose of this study is to assess whether tear secretion in patients with Parkinson's disease will be altered to exhibit a characteristic or diagnostic biomarker profile, that will be reflected in changes in the protein composition of tear fluid, which can be measured relatively easily, cost-effectively, and non-invasively. Tear fluid samples will be collected from Parkinson's patients, and through biochemical assays, the profile of proteins in tears will be characterized and compared to that from control subjects. The profiles will be analyzed with respect to any differences between Parkinson's patients and control subjects. If differences appear, the levels of these potential biomarkers in Parkinson's patients will be compared to the severity of their disease.

ELIGIBILITY:
Inclusion Criteria:

* established Parkinson's Disease for at least 6 months
* Healthy controls without neurological illness

Exclusion Criteria:

* currently taking anti-cholinergic medication
* dementia
* have an exposure to neuroleptic medications other than Quetiapine or Clozapine in the 6 months prior to screening
* have an active eye infection or have had eye surgery within 3 months prior to screening
* control subjects will be excluded if they have a history of neurological disease
* PD subjects will be excluded if they have an atypical Parkinsonian syndrome

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit participants with Parkinson's disease and controls from the Parkinson's Disease and Movement Disorder Center at the University of Southern California (USC) and from the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Tear protein composition to discriminate between participants with Parkinson's disease and healthy controls | up to 12 months
  4 potential biomarkers will be evaluated in collected tear fluid and will be followed longitudinally for 3-4 visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Hamm-Alvarez SF, Janga SR, Edman MC, Feigenbaum D, Freire D, Mack WJ, Okamoto CT, Lew MF. Levels of oligomeric alpha-Synuclein in reflex tears distinguish Parkinson's disease patients from healthy controls. Biomark Med. 2019 Dec;13(17):1447-1457. doi: 10.2217/bmm-2019-0315. Epub 2019 Sep 25. PMID 31552762